CLINICAL TRIAL: NCT02717208
Title: A Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Safety, Local Tolerability and Pharmacokinetic Characteristics After Administration of Eye-drop HL036 in Healthy Korean Male Volunteers (Phase I)
Brief Title: Phase 1 Study for Safety and Tolerability of HL036
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HanAll BioPharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HTR15I_1
Record Dates: First submitted 2016-02-18; First posted 2016-03-23 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-02

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- HL036 0.5mg/ml (Active Comparator): Administration : 2 times per day for one day
  Interventions: Biological: HL036; Biological: Vehicle
- HL036 5mg/ml (Active Comparator): Administration : 2 times per day for one day
  Interventions: Biological: HL036; Biological: Vehicle

INTERVENTIONS:
Biological: HL036
Biological: Vehicle

SUMMARY:
To evaluate the safety, local tolerability and pharmacokinetic characteristics after administration of eye-drop HL036 in healthy Korean male volunteers

DETAILED DESCRIPTION:
A total of 10 subjects will be dosed in each group with subjects randomized 8:2 to HL036 or placebo. Three of 10 subjects will be randomized to the sentinel dosing in each group. A safety data review as masking will be performed for 3days prior to the other subjects treatment. Treatment of high dose will proceed following a review of safety data from low dose.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who listened to the description about characteristics of this clinical trial and signed the IRB approved consent form before the whole screening tests
* Healthy Korean males volunteers who are 20 to 50 years old at screening procedure

Exclusion Criteria:

- Subjects who have a history of tuberculosis or have a positive Quantiferon Test

* Subjects who have treated live vaccine within 8 weeks prior to the first day of dosing or have a plan to treat it before the end of study
* Subjects who have presence or history of significant hepatic(including hepatitis B or C) , renal, neurological, immunological, respiratory , endocrine or hemato•oncology, cardiovascular, psychiatric disease
* Subjects who have presence or history of ophthalmological examination by the following

  ① History of ocular disease including keratitis, uveitis, retinitis, dry eye, strabismus or had suspected symptoms or signs

  ② Subjects who are under 20/40 of corrected visual acuity at screening

  ③ Subjects with a history of ocular surgery ( including subjects who had laser surgery in the previous 6 month from screening)

  ④ Subjects who had contact lens wear within 1 month or had side effects after wearing, unwilling to discontinue wear during the study period

  ⑤ Abnormalities following other ophthalmological examination
* Subjects who have a history of allergy to anti-TNF drug(infliximab, adalimumab, etanercept) or any similar product
* Subjects who had a history of drug abuse or a positive of drug abuse at urine test
* Subjects who have taken any prescribed drugs, herbal agents within 2 weeks or who have taken any over-the-counter (OTC) drugs including artificial tears or vitamins within 1 week prior to the first day of dosing (Investigators will determine his eligibility by considering the effect of the drug on his safety or pharmacokinetic results in case other inclusion/exclusion criteria is satisfied.)
* Subjects who have participated in another clinical trial or bioequivalence research with an IP within 3 months prior to the first day of dosing.
* Subjects who donated whole blood within 2 months or component blood within 1 month or who are donated within 1 month prior to the first day of dosing.
* Subjects who have currently drinks in excess of 21 units per week(1 unit = 10 g of pure alcohol) or would not be able to stop drinking alcohol during the study
* Subjects who have smoked in the 6 months or has used nicotine product or would not be able to stop smoking during the hospitalization Subjects who planned pregnancy or cannot use established contraceptions (e.g. infertility operation of the subject or partner, intrauterine contraceptive device of the partner, barrier contraception, diaphragm or condom use in combination during the test
* Subject who are judged as inappropriate for participating in the clinical trial by researcher because of causes including the test result of clinical laboratory

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 1 week

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 24 hours
Area under the plasma concentration versus time curve (AUC) | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital,Clinical Trial Center/ Clinical Research Institute, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided